CLINICAL TRIAL: NCT07159958
Title: The Effect of Simulation Supported Vulva Cancer and Vulva Self-Examination Training on Knowledge, Skills and Attitude Towards Clinical Practices: A Randomized Controlled Study
Brief Title: Simulation Supported Vulva Cancer and Self-Examination on Knowledge, Skills and Attitude
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Burcu KUCUKKAYA, Assoc. Prof., Trakya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2025-SBB-0332
Record Dates: First submitted 2025-08-30; First posted 2025-09-08 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Vulva Cancer; Nurse Role
Keywords: Simulation Supported Education; Vulva Self-Examination; Attitude Towards Clinical Practices
MeSH Terms: conditions — Vulvar Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training group (Experimental)
  Interventions: Other: Simulation-Based Vulvar Cancer and Self-Vulvar Examination Training
- Control group (No Intervention)

INTERVENTIONS:
Other: Simulation-Based Vulvar Cancer and Self-Vulvar Examination Training — The topics covered include the definition of vulvar cancer, risk factors, symptoms, preventive measures to protect against cancer, the definition of KKVM, and the steps involved in performing an examination. The inspection phase of the examination was demonstrated using a light source and mirror on a simulated model of the external genitalia. In addition, the topic was reiterated by explaining on the model how palpation examination is performed, when it should be performed, what signs and symptoms to look for, and in which cases a doctor should be consulted.
  Arms: Training group

SUMMARY:
Objective: The aim of this study was to examine the effect of simulation-assisted vulvar cancer and vulva self-examination training on knowledge, skills and attitudes towards clinical practices.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older,
* Able to read and write Turkish,
* Has not taken a course/seminar on vulvar cancer and self-vulvar examination,
* Enrolled in the Nursing Department of the Faculty of Health Sciences at Bartın University,
* Receiving education during the time period when the study is conducted,
* Volunteering to participate in the study.

Exclusion Criteria:

* Those who withdrew or dropped out of the study early,
* Those who were not willing to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2025-05-08 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-09-05 (Actual)

PRIMARY OUTCOMES:
Self-Vulva Examination Knowledge Level Form | change from before implamentation patent and after 1st and 4th weeks of practice
  The scale was developed by Karaman to assess knowledge and skills related to self-vulva examination. The KKVM Knowledge Form was created based on a review of studies in the field of vulvar cancer. It consists of 20 items for use in the form. The KKVM Knowledge Level Form consists of "Yes," "No," and "I don't know" options for participants to answer each item.
Attitude Scale Toward Clinical Practice for Nursing Students | change from before implamentation patent and after 1st and 4th weeks of practice
  The scale consists of 26 items and 4 subscales (Beliefs and Expectations Regarding Clinical Practice, Positive Approach to Clinical Practice, Negative Approach to Clinical Practice, and Personal Development) and is a 5-point Likert scale. The first sub-dimension has eight items, the second sub-dimension has seven items, the third sub-dimension has seven items, and the fourth sub-dimension has four items.
Self-Vulva Examination Skill Checklist Steps | change from before implamentation patent and after 1st and 4th weeks of practice
  Self-Vulva Examination Skill Checklist Steps

CONTACTS AND LOCATIONS:
Locations (1):
- Eskişehir Osmangazi University, Eskişehir, Turkey (Türkiye)